CLINICAL TRIAL: NCT03752281
Title: Long Term Social Assistance Receipt - An Observational Study of Health, Function, and Activity
Brief Title: Long Term Social Assistance Recipient in South Eastern Sweden - a Description of Health, Function, and Activity
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Linkoeping University (Other Government)
Collaborators: Linkoeping Municipality (Unknown)
Responsible Party: Principal Investigator, Bjorn Gerdle, Professor, Linkoeping University
Other Study IDs: TU-001-1811
Record Dates: First submitted 2018-11-19; First posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Vocational Rehabilitation
Keywords: Health, activity, function and long-term social assistance
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health and activity: The cohort consists of long-term social assistance recipients where there is need to investigate the health status and working ability.
  Interventions: Other: Investigation of health and activity

INTERVENTIONS:
Other: Investigation of health and activity — During a six months multidisciplinary investigation of health status, activity and working ability for individuals receiving long-term social assistance, the health and activity status as well as function will be described using established questionnaires and the International Classification of Functioning

SUMMARY:
There is a group of social assistance recipients which have difficulties in entering the labor market and thus remains in a long-term dependency on social assistance. More knowledge about individuals receiving long-term social assistance is needed in order to improve into work interventions for this group. Therefore, this study aims to describe variables of health, function and activity in participants receiving long-term social assistance.

DETAILED DESCRIPTION:
There is a group of social assistance recipients who have difficulties in entering the labor market and thus remains in a long-term dependency on social assistance. More knowledge about individuals receiving long-term social assistance is needed in order to improve into-work interventions for this group. Therefore, this study aims to describe variables of health, function and activity in participants receiving long-term social assistance. Individuals who have received social assistance during more than three years, who report physical and/or psychological difficulties, and/or have a complex social situation will be asked for participation in a six months activity-based investigation including contact with social worker, psychologist, occupational therapist, physical therapist and labor market consultant. The intervention aims to clarify the participants hinders and resources for entering the labor market. The participants are going to answer a questionnaire about health, function, and activity before and after the investigation. In addition, the participants function and ability to perform activities will be classified using the International Classification of Functioning (ICF). Data from the questionnaires and from ICF recordings will be used to describe variables of health, function and ability to be active. Participants who manage to get closer to, or enter into, the labor market will be asked to participate in a qualitative interview study about the experiences of the change. In addition, social workers will be asked to participate in focus-group interviews about experiences from the professional contact and work with the participants. The quantitative data will be analysed using traditional statistics and multivariate data analysis. Qualitative data will be analysed using qualitative content analysis.

ELIGIBILITY:
Inclusion Criteria:

* Long-term social assistance recipient (more than three years)
* Putative ill-health (physical, psychological and/or social)
* No present plan how to reach the labor market
* Need of clarifying the working ability

Exclusion Criteria:

* Homelessness
* Severe psychiatric illness
* Abuse of alcohol or substances

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who have been social assistance recipients for at least three years and who not have a plan how to get closer to the labor market. There may be signs of different kinds of ill-health such as physical, pshychological and/or social ill-health. The social worker responsible for decision about the monetary support identifies a need for establishing the working ability of the individual with the aim to agree on a plan towards self-sufficiency.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life | Change between the beginning and the end of the six months intervention
  The change in participants self-rated experience of quality of life is going to be described using EuroQol 5 Dimensions which contains a rating of the ability to perform activities, and also a score of the total quality of life experience.
Change in self-rated function and ability to be active | Change between the beginning and the end of the six months intervention
  The change in participants self-rated function and ability to be active is going to be described using the World Health Organisation Disability Assessment Schedule (WHODAS) which contains five-grade ratings of factors including functioning, activity and participation.
Change in objective description of function and ability to be active | Change between the beginning and the end of the six months intervention
  The change in an objective classification of function, activity, participation and environmental factors affecting disability will be described according to the International Classification of Functioning (ICF) in the beginning and at the end of the six month intervention. The ICF contains a number of components, where each component can be scored using a five-grade scale to clarify the magnitude of disability.

SECONDARY OUTCOMES:
Qualitative description of experiences about an increase in activity ability | After the six moths intervention
  Participants experiences about a change towards higher ability to be active will be described using qualitative interviews.
Qualitative description of social workers experiences from the work with long-term social assistance recipients | After the six moths intervention
  Social workers experiences from their work with helping clients to get closer to the labor market will be described using qualitative interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Linn Karlsson, PhD, Study Chair — Linkoeping Municipality, Linkoeping University
Locations (1):
- Faculty of Health Sciences, Linköping University, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The co-authors will have access to the underlying interview data for the qualitative analysis. Quantitative data will be coded and not able to identify to any participant for the co-authors. However, it may be necessary for the co-authors to get access to the quantitative (anonymized) raw data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available during analysis and manuscript writing. Probable for about six moths per paper.
Access Criteria: Co-authors who will be participating in analysis and manuscript preparation.

REFERENCES:
- [Background] van Vilsteren M, van Oostrom SH, de Vet HC, Franche RL, Boot CR, Anema JR. Workplace interventions to prevent work disability in workers on sick leave. Cochrane Database Syst Rev. 2015 Oct 5;2015(10):CD006955. doi: 10.1002/14651858.CD006955.pub3. PMID 26436959
- [Background] Vogel N, Schandelmaier S, Zumbrunn T, Ebrahim S, de Boer WE, Busse JW, Kunz R. Return-to-work coordination programmes for improving return to work in workers on sick leave. Cochrane Database Syst Rev. 2017 Mar 30;3(3):CD011618. doi: 10.1002/14651858.CD011618.pub2. PMID 28358173
- [Background] Arends I, Bruinvels DJ, Rebergen DS, Nieuwenhuijsen K, Madan I, Neumeyer-Gromen A, Bultmann U, Verbeek JH. Interventions to facilitate return to work in adults with adjustment disorders. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD006389. doi: 10.1002/14651858.CD006389.pub2. PMID 23235630
- [Background] Madden RH, Dune T, Lukersmith S, Hartley S, Kuipers P, Gargett A, Llewellyn G. The relevance of the International Classification of Functioning, Disability and Health (ICF) in monitoring and evaluating Community-based Rehabilitation (CBR). Disabil Rehabil. 2014;36(10):826-37. doi: 10.3109/09638288.2013.821182. Epub 2013 Aug 14. PMID 23944180
- [Background] Prodinger B, Stucki G, Coenen M, Tennant A. The measurement of functioning using the International Classification of Functioning, Disability and Health: comparing qualifier ratings with existing health status instruments. Disabil Rehabil. 2019 Mar;41(5):541-548. doi: 10.1080/09638288.2017.1381186. Epub 2017 Oct 8. PMID 28988490
- See also: The national board of health and welfare in Sweden — http://www.socialstyrelsen.se/
- See also: The social service act — http://www.riksdagen.se/sv/dokument-lagar/dokument/svensk-forfattningssamling/socialtjanstlag-2001453_sfs-2001-453